CLINICAL TRIAL: NCT05909787
Title: Prevalence of Oral Disorders in Children Identified by Parents in the Context of ENT Pathologies
Brief Title: Prevalence of Oral Disorders in Children in ENT Pathologies
Acronym: Preora
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APHP230191; IDRCB: 2023-A00201-44 (Registry Identifier: French Health Authority)
Record Dates: First submitted 2023-06-09; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-04

CONDITIONS: Eating Disorders; Language Disorders
Keywords: Eating disorders; Language disorders; Childhood
MeSH Terms: conditions — Feeding and Eating Disorders; Language Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Auto-questionnaire MCH (Montreal Children's Hospital) (Experimental): Auto-questionnaire MCH (Montreal Children's Hospital)
  Interventions: Other: Auto-questionnaire

INTERVENTIONS:
Other: Auto-questionnaire — MCH (Montreal Children's Hospital) self questionnaire completed by the parents

SUMMARY:
Many children have eating and verbal oral disorders. Our research entitled: PREORA aims to study the prevalence of oral disorders presented in children consulting in ENT department for three months (n = 2000). This first study will be carried out by passing the MCH (Montreal Children's Hospital) feeding scale, a self-questionnaire completed by the parents, in order to assess the presence of disorders according to the parents and will allow us to present oral disorders (Score > 70).

DETAILED DESCRIPTION:
Over a period of inclusion of 3 months, the doctors of the departement ONT, Robert Debré Hospital, will give written and oral information to the holders of parental authority and to the child at the beginning of the consultation. After a 15-minute reflection period (consultation time), if they agree to participate, parents will answer the doctor's questions and then complete the self-questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Patients consulting at ENT departement Robert Debré Hospital
* Age 0-17 years
* Parents and children informed and given their oral consent for the study and speaking french

Exclusion Criteria:

* Refusal of parents/children to participate

Ages: 1 Day to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2000 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Difficulty in feeding | 50 minutes
  MCH self questionnaire / HME score

CONTACTS AND LOCATIONS:
Overall Officials: Natacha TEISSIER, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris

IPD SHARING:
Plan to Share IPD: No